CLINICAL TRIAL: NCT04517669
Title: A Non-Interventional Multinational Study of Tofacitinib in Patients Treated for Psoriatic Arthritis
Brief Title: Effectiveness of Treatment With Tofacitinib in Patients With Psoriatic Arthritis in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921332; TOPSATI (Other: Alias Study Number)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a Multinational Study of Tofacitinib in Patients Treated for Psoriatic Arthritis in order to evaluate the effectiveness of treatment with tofacitinib on disease activity, remission, and Quality of Life, in a real-world setting over a 12-month observation period

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Patients aged ≥ 18 years
2. Moderate to severe PsA disease activity diagnosed
3. Patients for whom the physician's decision has been made to initiate treatment with tofacitinib, in usual clinical practice conditions and in compliance with the local label
4. Patients are treatment naïve to tofacitinib on the date of providing informed consent
5. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study
6. Patients on DMARDs must have not had a treatment change in the past 3 months

Exclusion Criteria: Patients meeting any of the following criteria will not be included in the study:

1. Contraindications according to the Xeljanz® (tofacitinib) Prescribing Information
2. Receipt of any investigational drug within 3 months before study inclusion
3. Patient is pregnant or breastfeeding
4. Recent herpes zoster infection (within past 6 months) or history of severe disseminated herpes zoster infection
5. Active treatment for a malignancy
6. Concomitant treatment with a biological disease-modifying antirheumatic drugs (bDMARD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll approximately 500 patients from rheumatologists and/or PsA specialist centers in 10 countries (Belgium, Czech Republic, Denmark, Finland, France, Israel, Netherlands, Spain, Sweden, and Switzerland) over an enrollment period of 12 months. The above list of countries are anticipated to participate in this study, however additional countries may be included at a later time. Each patient will have up to 12 months of follow-up for a total study duration of 24 months. Consecutive patients attending a routine clinical visit will be invited to participate if they meet the eligibility criteria for the study and are to start on treatment with tofacitinib for active PsA.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- Belgium (3):
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - AZ Sint-Jan, Bruges
  - Nova Reuma Społka Partnerska, Genk
- Sygehus Vendsyssel Hospital, Hjørring, Denmark
- Turku University Hospital, Turku, Finland
- France (8):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier Jean Rougier, Cahors
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand
  - Hopital Pasteur, Nice
  - CHR Orleans, Orléans
  - Hopital Purpan, Toulouse
  - CHU Tours - Hôpital Trousseau, Tours
- Israel (12):
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Rambam Health Care Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Hadassah Hebrew University Medical Center - Ein Kerem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Baruch Padeh Medical Center - Poriya, Tiberias
- Netherlands (2):
  - Medisch Spectrum Twente, Haaksbergerstraat, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
- Spain (10):
  - C.H. Universitario de Vigo- Hospital Meixoeiro, Vigo, Galicia
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital de Especialidades de Jerez de la Frontera, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Quironsalud Infanta Luisa, Seville
- Sweden (4):
  - Lund University, Lund
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Karolinska University Hospital, Solna, Stockholm
  - Norrlands University Hospital Umeå, Reumatologiska kliniken Västerbotten, Umeå

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with psoriatic arthritis (PsA) and treated with tofacitinib in routine clinical practice were included in this prospective study.
Pre-assignment Details: A total of 116 participants from rheumatologists and/or PsA specialist centres across 8 countries (Belgium, Denmark, Finland, France, Israel, Netherlands, Spain, and Sweden) signed the informed consent.
Groups:
- All Participants: Participants diagnosed with PsA and treated with tofacitinib in routine clinical practice were included. No study drug was administered as part of this study. Participants were followed for up to 12 months.
Period: Overall Study
Arm/Group | All Participants
Started | 116
Safety (Started Tofacitinib Irrespective of Eligibility Criteria) | 113
Full Analysis Set | 109
Completed | 59
Not Completed | 57
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Drug withdrawn | 44
Not completed — Other | 1
Not completed — Eligibility criteria not met | 4
Not completed — Did not receive treatment | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who received at least one dose (including partial dose) of study medication independently of inclusion/exclusion criteria.
Arm/Group | All Participants
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Low Disease Activity (LDA) Based on Psoriatic Arthritis Disease Activity Score (PASDAS) at Month 6
Description: PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global psoriatic arthritis assessment (PAA), physician global PAA, each scored on 100 mm visual analog scale (VAS), 0=no disease activity (DA), 100=maximum DA; tender joint count (TJC) (0-68); swollen joint count (SJC) (0-66); Leed's Enthesitis index (LEI) score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; physical component summary (PCS) of short form 36 (SF-36) score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and C-reactive protein (CRP) in milligram per liter (mg/L). PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease. LDA was defined as PASDAS score less than or equal to (<=) 3.2.
Time Frame: At Month 6
Population: Full analysis set (FAS) included all enrolled participants who received at least one dose (including partial dose) of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
Percentage of participants
  Overall | 43.1 [29.9 to 56.3]
  Tofacitinib monotherapy: number analyzed (Participants) | 54
  Tofacitinib monotherapy | 46.9 [31.4 to 62.4]
  Combined tofacitinib and methotrexate (MTX) therapy: number analyzed (Participants) | 17
  Combined tofacitinib and methotrexate (MTX) therapy | 33.4 [9.4 to 57.5]
  Combined tofacitinib and other conventional synthetic disease-modifying antirheumatic drug (csDMARD): number analyzed (Participants) | 1
  Combined tofacitinib and other conventional synthetic disease-modifying antirheumatic drug (csDMARD) | 4.0 [NA to NA] — Upper limit and lower limit of 95% confidence interval (CI) could not be calculated due to insufficient number of participants with events.

2. Secondary Outcome: Percentage of Participants Who Achieved LDA Based on PASDAS at Months 3 and 12
Description: PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease. LDA was defined as PASDAS score less than or equal to (<=) 3.2.
Time Frame: At Month 3 and Month 12
Population: The FAS included all enrolled participants who received at least one dose (including partial dose) of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Percentage of participants
  Overall-Month 3 | 23.5 [13.9 to 36.9]
  Tofacitinib monotherapy-Month 3: number analyzed (Participants) | 38
  Tofacitinib monotherapy-Month 3 | 21.1 [10.8 to 36.6]
  Combined tofacitinib and MTX therapy-Month 3: number analyzed (Participants) | 12
  Combined tofacitinib and MTX therapy-Month 3 | 33.3 [13.6 to 61.2]
  Combined tofacitinib and other csDMARD-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 3 | 0 [0.0 to 82.9]
  Overall-Month 12: number analyzed (Participants) | 26
  Overall-Month 12 | 46.2 [28.7 to 64.5]
  Tofacitinib monotherapy-Month 12: number analyzed (Participants) | 19
  Tofacitinib monotherapy-Month 12 | 47.4 [27.3 to 68.3]
  Combined tofacitinib and MTX therapy-Month 12: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy-Month 12 | 42.9 [15.8 to 75.0]
  Combined tofacitinib and other csDMARD-Month 12: number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Who Achieved Minimum Disease Activity (MDA) at Months 3, 6 and 12
Description: A participant was classified as MDA achieved if they met 5 of 7 criteria: (i) (TJC66) <=1, (ii) (SJC68)<=1, (iii) psoriasis area and severity index (PASI) score <=1 (PASI=combined assessment of lesion severity and area affected into single score; range=0 [no disease] to 72 [maximal disease], higher scores=more disease. or body surface area (BSA) <=3%,(iv) patient pain assessment (VAS, 0-100) <=15; where 0='no pain' and 100='pain as severe as can be imagined', higher scores=more pain, (v) patient global assessment (VAS, 0-100) <=20, where 0='lowest level of disease activity' and 100= 'highest level of disease activity, higher scores=more disease activity, (vi) health assessment questionnaire-disability index (HAQ- DI) <=0.5; scale ranged=0-3, where 0='normal or no difficulty' and 3='inability to perform', higher scores=more difficulty, (vii) tender enthesial points <=1 using Leed's index range=0=non tender to 6=more enthesitis burden, higher scores=more burden.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 91
Percentage of participants
  Overall-Month 3 | 17.6 [11.0 to 26.8]
  Tofacitinib monotherapy-Month 3: number analyzed (Participants) | 66
  Tofacitinib monotherapy-Month 3 | 16.7 [9.4 to 27.6]
  Combined tofacitinib and MTX therapy-Month 3: number analyzed (Participants) | 23
  Combined tofacitinib and MTX therapy-Month 3 | 21.7 [9.2 to 42.3]
  Combined tofacitinib and other csDMARD-Month 3: number analyzed (Participants) | 2
  Combined tofacitinib and other csDMARD-Month 3 | 0 [0.0 to 71.1]
  Overall-Month 6: number analyzed (Participants) | 71
  Overall-Month 6 | 42.3 [31.4 to 53.9]
  Tofacitinib monotherapy-Month 6: number analyzed (Participants) | 50
  Tofacitinib monotherapy-Month 6 | 42.0 [29.4 to 55.8]
  Combined tofacitinib and MTX therapy-Month 6: number analyzed (Participants) | 20
  Combined tofacitinib and MTX therapy-Month 6 | 45.0 [25.8 to 65.8]
  Combined tofacitinib and other csDMARD-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 6 | 0 [0.0 to 82.9]
  Overall-Month 12: number analyzed (Participants) | 57
  Overall-Month 12 | 43.9 [31.8 to 56.7]
  Tofacitinib monotherapy-Month 12: number analyzed (Participants) | 40
  Tofacitinib monotherapy-Month 12 | 45.0 [30.7 to 60.2]
  Combined tofacitinib and MTX therapy-Month 12: number analyzed (Participants) | 16
  Combined tofacitinib and MTX therapy-Month 12 | 43.8 [23.1 to 66.8]
  Combined tofacitinib and other csDMARD-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 12 | 0 [0.0 to 82.9]

4. Secondary Outcome: Percentage of Participants Who Achieved Remission Based on PASDAS at Months 3, 6 and 12
Description: PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease. Remission was defined as PASDAS score less than or equal to (<=) 1.9.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 66
Percentage of participants
  Overall-Month 3 | 12.1 [6.0 to 22.4]
  Tofacitinib monotherapy-Month 3: number analyzed (Participants) | 49
  Tofacitinib monotherapy-Month 3 | 14.3 [6.8 to 27.0]
  Combined tofacitinib and MTX therapy-Month 3: number analyzed (Participants) | 14
  Combined tofacitinib and MTX therapy-Month 3 | 7.1 [0.0 to 33.5]
  Combined tofacitinib and other csDMARD-Month 3: number analyzed (Participants) | 3
  Combined tofacitinib and other csDMARD-Month 3 | 0 [0.0 to 62.0]
  Overall-Month 6: number analyzed (Participants) | 51
  Overall-Month 6 | 15.7 [7.9 to 28.3]
  Tofacitinib monotherapy-Month 6: number analyzed (Participants) | 35
  Tofacitinib monotherapy-Month 6 | 20.0 [9.7 to 36.2]
  Combined tofacitinib and MTX therapy-Month 6: number analyzed (Participants) | 15
  Combined tofacitinib and MTX therapy-Month 6 | 6.7 [0.0 to 31.8]
  Combined tofacitinib and other csDMARD-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 6 | 0 [0.0 to 82.9]
  Overall-Month 12: number analyzed (Participants) | 37
  Overall-Month 12 | 21.6 [11.1 to 37.4]
  Tofacitinib monotherapy-Month 12: number analyzed (Participants) | 27
  Tofacitinib monotherapy-Month 12 | 25.9 [12.9 to 44.9]
  Combined tofacitinib and MTX therapy-Month 12: number analyzed (Participants) | 9
  Combined tofacitinib and MTX therapy-Month 12 | 11.1 [0.0 to 45.7]
  Combined tofacitinib and other csDMARD-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 12 | 0 [0.0 to 82.9]

5. Secondary Outcome: Percentage of Participants Who Achieved Remission Based on Disease Activity in Psoriatic Arthritis (DAPSA) Score at Months 3, 6 and 12
Description: DAPSA was composite disease activity measure and was calculated as: SJC66 + TJC68 + patient global assessment VAS (0 to 10 cm VAS, 0= excellent and 10= poor, higher scores indicated more disease activity) + patient pain assessment (0 to 10 cm VAS, 0= no pain, 10= worst possible pain, higher scores indicated more pain) + CRP (mg/dL). DAPSA score ranged from 0 to 164, higher scores indicated more disease activity. Remission was defined as DAPSA score =<4.0.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 53
Percentage of participants
  Overall-Month 3 | 11.3 [4.9 to 22.9]
  Tofacitinib monotherapy-Month 3: number analyzed (Participants) | 43
  Tofacitinib monotherapy-Month 3 | 11.6 [4.6 to 24.9]
  Combined tofacitinib and MTX therapy-Month 3: number analyzed (Participants) | 9
  Combined tofacitinib and MTX therapy-Month 3 | 11.1 [0.0 to 45.7]
  Combined tofacitinib and other csDMARD-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 3 | 0 [0.0 to 82.9]
  Overall-Month 6: number analyzed (Participants) | 45
  Overall-Month 6 | 28.9 [17.6 to 43.5]
  Tofacitinib monotherapy-Month 6: number analyzed (Participants) | 33
  Tofacitinib monotherapy-Month 6 | 36.4 [22.1 to 53.4]
  Combined tofacitinib and MTX therapy-Month 6: number analyzed (Participants) | 12
  Combined tofacitinib and MTX therapy-Month 6 | 8.3 [0.0 to 37.5]
  Combined tofacitinib and other csDMARD-Month 6: number analyzed (Participants) | 0
  Overall-Month 12: number analyzed (Participants) | 31
  Overall-Month 12 | 38.7 [23.7 to 56.2]
  Tofacitinib monotherapy-Month 12: number analyzed (Participants) | 21
  Tofacitinib monotherapy-Month 12 | 47.6 [28.3 to 67.6]
  Combined tofacitinib and MTX therapy-Month 12: number analyzed (Participants) | 10
  Combined tofacitinib and MTX therapy-Month 12 | 20.0 [4.6 to 52.1]
  Combined tofacitinib and other csDMARD-Month 12: number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Impact of Disease 12 Questions (PsAID12) Score at Months 3, 6 and 12
Description: PsAID12: questionnaire used for evaluating how much PsA impacted quality of life (QoL) and comprised of following domains: Pain, Fatigue, Skin problems, Work and/or leisure activities, Function, Discomfort, Sleep disturbance, Coping, Anxiety, Embarrassment, Social life and Depression. Each one of domain was based on a 0-10 numerical rating scale (NRS) and with different weight. PsAID12= (PsAID12.Q1 [pain] NRS value*3) +(PsAID12.Q2[fatigue] NRS value*2) +(PsAID12.Q3 [skin] NRS value*2) +(PsAID12.Q4[Work and/or leisure activities] NRS value*2) +(PsAID12.Q5[function] NRS value*2) +(PsAID12.Q6[discomfort]NRS value*2) +(PsAID12.Q7[sleep] NRS value*2) +(PsAID12.Q8 [coping]NRS value*1) +(PsAID12.Q9[anxiety] NRS value*1) +(PsAID12.Q10[embarrassment] NRS value*1) +(PsAID12.Q11[social life] NRS value*1) +(PsAID12.Q12[depression] NRS value*1). Total is divided by 20 for final score. Range of final PsAID score is 0-10 (higher numbers indicate worse status).
Time Frame: Baseline (measurement at enrollment), at Month 3, Month 6 and Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 89
Units on a scale
  Overall-Month 3 | -1.3 [-1.69 to -0.84]
  Tofacitinib monotherapy-Month 3: number analyzed (Participants) | 65
  Tofacitinib monotherapy-Month 3 | -1.4 [-1.91 to -0.86]
  Combined tofacitinib and MTX therapy-Month 3: number analyzed (Participants) | 21
  Combined tofacitinib and MTX therapy-Month 3 | -1.0 [-1.84 to -0.15]
  Combined tofacitinib and other csDMARD-Month 3: number analyzed (Participants) | 3
  Combined tofacitinib and other csDMARD-Month 3 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Overall-Month 6: number analyzed (Participants) | 69
  Overall-Month 6 | -1.3 [-1.79 to -0.80]
  Tofacitinib monotherapy-Month 6: number analyzed (Participants) | 49
  Tofacitinib monotherapy-Month 6 | -1.5 [-2.06 to -0.87]
  Combined tofacitinib and MTX therapy-Month 6: number analyzed (Participants) | 19
  Combined tofacitinib and MTX therapy-Month 6 | -0.9 [-1.91 to 0.08]
  Combined tofacitinib and other csDMARD-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 6 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Overall-Month 12: number analyzed (Participants) | 58
  Overall-Month 12 | -1.1 [-1.61 to -0.56]
  Tofacitinib monotherapy-Month 12: number analyzed (Participants) | 41
  Tofacitinib monotherapy-Month 12 | -1.3 [-1.94 to -0.64]
  Combined tofacitinib and MTX therapy-Month 12: number analyzed (Participants) | 16
  Combined tofacitinib and MTX therapy-Month 12 | -0.7 [-1.69 to 0.25]
  Combined tofacitinib and other csDMARD-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 12 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.

7. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC-EI) Score at Months 3, 6 and 12
Description: The SPARCC-EI evaluated 16 enthesial sites: greater trochanter (Right/Left [R/L]), quadriceps tendon insertion into the patella (R/L), patellar ligament insertion into the patella and tibial tuberosity (R/L), achilles tendon insertion (R/L), plantar fascia insertion (R/L), medial epicondyles (R/L), lateral epicondyles (R/L) and supraspinatus insertion (R/L) for the presence or absence of tenderness. Tenderness at each site was quantified as: 0 = non-tender and 1 = tender. The maximum score of the SPARCC-EI was 16. SPARCC-EI score range: 0 (no enthesitis) to 16 (enthesitis is present at all assessed sites), higher scores indicated more presence of enthesitis.
Time Frame: Baseline (measurement at enrollment), at Month 3, Month 6 and Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 57
Units on a scale
  Overall-Month 3 | 0.1 [-0.67 to 0.85]
  Tofacitinib monotherapy-Month 3: number analyzed (Participants) | 40
  Tofacitinib monotherapy-Month 3 | 0.1 [-0.80 to 0.95]
  Combined tofacitinib and MTX therapy-Month 3: number analyzed (Participants) | 15
  Combined tofacitinib and MTX therapy-Month 3 | 0.2 [-1.87 to 2.18]
  Combined tofacitinib and other csDMARD-Month 3: number analyzed (Participants) | 2
  Combined tofacitinib and other csDMARD-Month 3 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Overall-Month 6: number analyzed (Participants) | 45
  Overall-Month 6 | -0.8 [-1.47 to -0.21]
  Tofacitinib monotherapy-Month 6: number analyzed (Participants) | 32
  Tofacitinib monotherapy-Month 6 | -0.4 [-1.17 to 0.28]
  Combined tofacitinib and MTX therapy-Month 6: number analyzed (Participants) | 13
  Combined tofacitinib and MTX therapy-Month 6 | -1.8 [-3.20 to -0.39]
  Combined tofacitinib and other csDMARD-Month 6: number analyzed (Participants) | 0
  Overall-Month 12: number analyzed (Participants) | 36
  Overall-Month 12 | -0.3 [-0.95 to 0.44]
  Tofacitinib monotherapy-Month 12: number analyzed (Participants) | 24
  Tofacitinib monotherapy-Month 12 | 0.0 [-0.81 to 0.82]
  Combined tofacitinib and MTX therapy-Month 12: number analyzed (Participants) | 12
  Combined tofacitinib and MTX therapy-Month 12 | -0.9 [-2.42 to 0.71]
  Combined tofacitinib and other csDMARD-Month 12: number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants Who Achieved LDA According to Body Mass Index (BMI) at Months 3, 6 and 12
Description: BMI = Weight (kilograms [kg]) / Height (meter square [m]^2). LDA was defined as PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease. In this outcome measure, participants with PASDAS scores are reported according to BMI categories of 18.5 - <25 kg/m^2, 25 - <30 kg/m^2, >= 30 kg/m^2 and missing.
Time Frame: At Month 3, Month 6 and Month 12
Population: The FAS included all enrolled participants who received at least one dose (including partial dose) of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows. All participants in "Overall Number of Participants Analyzed" contributed data to the table but may not have data evaluable for every row.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: 18.5 - <25 kg/m^2-Month 3: number analyzed (Participants) | 10
  Overall: 18.5 - <25 kg/m^2-Month 3 | 2
  Overall: 25 - <30 kg/m^2-Month 3: number analyzed (Participants) | 20
  Overall: 25 - <30 kg/m^2-Month 3 | 6
  Overall: >= 30 kg/m^2-Month 3: number analyzed (Participants) | 18
  Overall: >= 30 kg/m^2-Month 3 | 3
  Overall: Missing-Month 3: number analyzed (Participants) | 3
  Overall: Missing-Month 3 | 1
  Overall: 18.5 - <25 kg/m^2-Month 6: number analyzed (Participants) | 12
  Overall: 18.5 - <25 kg/m^2-Month 6 | 8
  Overall: 25 - <30 kg/m^2-Month 6: number analyzed (Participants) | 15
  Overall: 25 - <30 kg/m^2-Month 6 | 8
  Overall: >= 30 kg/m^2-Month 6: number analyzed (Participants) | 8
  Overall: >= 30 kg/m^2-Month 6 | 2
  Overall: Missing-Month 6: number analyzed (Participants) | 3
  Overall: Missing-Month 6 | 2
  Overall: 18.5 - <25 kg/m^2-Month 12: number analyzed (Participants) | 12
  Overall: 18.5 - <25 kg/m^2-Month 12 | 5
  Overall: 25 - <30 kg/m^2-Month 12: number analyzed (Participants) | 8
  Overall: 25 - <30 kg/m^2-Month 12 | 4
  Overall: >= 30 kg/m^2-Month 12: number analyzed (Participants) | 5
  Overall: >= 30 kg/m^2-Month 12 | 2
  Overall: Missing-Month 12: number analyzed (Participants) | 1
  Overall: Missing-Month 12 | 1
  Tofacitinib monotherapy: 18.5 - <25 kg/m^2-Month 3: number analyzed (Participants) | 6
  Tofacitinib monotherapy: 18.5 - <25 kg/m^2-Month 3 | 1
  Tofacitinib monotherapy: 25 - <30 kg/m^2-Month 3: number analyzed (Participants) | 18
  Tofacitinib monotherapy: 25 - <30 kg/m^2-Month 3 | 5
  Tofacitinib monotherapy: >= 30 kg/m^2-Month 3: number analyzed (Participants) | 12
  Tofacitinib monotherapy: >= 30 kg/m^2-Month 3 | 1
  Tofacitinib monotherapy: Missing-Month 3: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Missing-Month 3 | 1
  Tofacitinib monotherapy: 18.5 - <25 kg/m^2-Month 6: number analyzed (Participants) | 6
  Tofacitinib monotherapy: 18.5 - <25 kg/m^2-Month 6 | 4
  Tofacitinib monotherapy: 25 - <30 kg/m^2-Month 6: number analyzed (Participants) | 14
  Tofacitinib monotherapy: 25 - <30 kg/m^2-Month 6 | 8
  Tofacitinib monotherapy: >= 30 kg/m^2-Month 6: number analyzed (Participants) | 5
  Tofacitinib monotherapy: >= 30 kg/m^2-Month 6 | 1
  Tofacitinib monotherapy: Missing-Month 6: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Missing-Month 6 | 2
  Tofacitinib monotherapy: 18.5 - <25 kg/m^2-Month 12: number analyzed (Participants) | 7
  Tofacitinib monotherapy: 18.5 - <25 kg/m^2-Month 12 | 3
  Tofacitinib monotherapy: 25 - <30 kg/m^2-Month 12: number analyzed (Participants) | 8
  Tofacitinib monotherapy: 25 - <30 kg/m^2-Month 12 | 4
  Tofacitinib monotherapy: >= 30 kg/m^2-Month 12: number analyzed (Participants) | 3
  Tofacitinib monotherapy: >= 30 kg/m^2-Month 12 | 1
  Tofacitinib monotherapy: Missing-Month 12: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Missing-Month 12 | 1
  Combined tofacitinib and MTX therapy: 18.5 - <25 kg/m^2-Month 3: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: 18.5 - <25 kg/m^2-Month 3 | 1
  Combined tofacitinib and MTX therapy: 25 - <30 kg/m^2-Month 3: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: 25 - <30 kg/m^2-Month 3 | 1
  Combined tofacitinib and MTX therapy: >= 30 kg/m^2-Month 3: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: >= 30 kg/m^2-Month 3 | 2
  Combined tofacitinib and MTX therapy: Missing-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: Missing-Month 3 | 0
  Combined tofacitinib and MTX therapy: 18.5 - <25 kg/m^2-Month 6: number analyzed (Participants) | 6
  Combined tofacitinib and MTX therapy: 18.5 - <25 kg/m^2-Month 6 | 4
  Combined tofacitinib and MTX therapy: 25 - <30 kg/m^2-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: 25 - <30 kg/m^2-Month 6 | 0
  Combined tofacitinib and MTX therapy: >= 30 kg/m^2-Month 6: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: >= 30 kg/m^2-Month 6 | 1
  Combined tofacitinib and MTX therapy: Missing-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: Missing-Month 6 | 0
  Combined tofacitinib and MTX therapy: 18.5 - <25 kg/m^2-Month 12: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: 18.5 - <25 kg/m^2-Month 12 | 2
  Combined tofacitinib and MTX therapy: >= 30 kg/m^2-Month 12: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: >= 30 kg/m^2-Month 12 | 1
  Combined tofacitinib and other csDMARD: >= 30 kg/m^2-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: >= 30 kg/m^2-Month 3 | 0

9. Secondary Outcome: Number of Participants Who Achieved LDA According to Treatment Line at Months 3, 6 and 12
Description: Participants who achieved LDA according to treatment line were reported in this outcome measure. Treatment line included: tofacitinib monotherapy, combination therapy with MTX, and combination therapy with other csDMARDs. LDA was defined as PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: Tofacitinib as monotherapy-Month 3: number analyzed (Participants) | 38
  Overall: Tofacitinib as monotherapy-Month 3 | 8
  Overall: Combination therapy with MTX-Month 3: number analyzed (Participants) | 12
  Overall: Combination therapy with MTX-Month 3 | 4
  Overall: Combination with other csDMARD-Month 3: number analyzed (Participants) | 1
  Overall: Combination with other csDMARD-Month 3 | 0
  Overall: Tofacitinib as monotherapy-Month 6: number analyzed (Participants) | 27
  Overall: Tofacitinib as monotherapy-Month 6 | 15
  Overall: Combination therapy with MTX-Month 6: number analyzed (Participants) | 11
  Overall: Combination therapy with MTX-Month 6 | 5
  Overall: Tofacitinib as monotherapy-Month 12: number analyzed (Participants) | 19
  Overall: Tofacitinib as monotherapy-Month 12 | 9
  Overall: Combination therapy with MTX-Month 12: number analyzed (Participants) | 7
  Overall: Combination therapy with MTX-Month 12 | 3
  Tofacitinib monotherapy: Tofacitinib as monotherapy-Month 3: number analyzed (Participants) | 38
  Tofacitinib monotherapy: Tofacitinib as monotherapy-Month 3 | 8
  Tofacitinib monotherapy: Tofacitinib as monotherapy-Month 6: number analyzed (Participants) | 27
  Tofacitinib monotherapy: Tofacitinib as monotherapy-Month 6 | 15
  Tofacitinib monotherapy: Tofacitinib as monotherapy-Month 12: number analyzed (Participants) | 19
  Tofacitinib monotherapy: Tofacitinib as monotherapy-Month 12 | 9
  Combined tofacitinib and MTX therapy: Combination therapy with MTX-Month 3: number analyzed (Participants) | 12
  Combined tofacitinib and MTX therapy: Combination therapy with MTX-Month 3 | 4
  Combined tofacitinib and MTX therapy: Combination therapy with MTX-Month 6: number analyzed (Participants) | 11
  Combined tofacitinib and MTX therapy: Combination therapy with MTX-Month 6 | 5
  Combined tofacitinib and MTX therapy: Combination therapy with MTX-Month 12: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Combination therapy with MTX-Month 12 | 3
  Combined tofacitinib and other csDMARD: Combination with other csDMARD-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Combination with other csDMARD-Month 3 | 0

10. Secondary Outcome: Number of Participants Who Achieved LDA According to Duration of Current Episode Symptoms of at Least 6 Weeks Prior to Enrollment at Months 3, 6 and 12
Description: Duration of current episode of symptoms prior to enrollment were presented as: < 6, >=6 weeks. LDA was defined as PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: < 6 weeks-Month 3: number analyzed (Participants) | 17
  Overall: < 6 weeks-Month 3 | 4
  Overall: >= 6 weeks-Month 3: number analyzed (Participants) | 32
  Overall: >= 6 weeks-Month 3 | 6
  Overall: Missing-Month 3: number analyzed (Participants) | 2
  Overall: Missing-Month 3 | 2
  Overall: < 6 weeks-Month 6: number analyzed (Participants) | 19
  Overall: < 6 weeks-Month 6 | 11
  Overall: >= 6 weeks-Month 6: number analyzed (Participants) | 18
  Overall: >= 6 weeks-Month 6 | 8
  Overall: Missing-Month 6: number analyzed (Participants) | 1
  Overall: Missing-Month 6 | 1
  Overall: < 6 weeks-Month 12: number analyzed (Participants) | 14
  Overall: < 6 weeks-Month 12 | 4
  Overall: >= 6 weeks-Month 12: number analyzed (Participants) | 12
  Overall: >= 6 weeks-Month 12 | 8
  Tofacitinib monotherapy: < 6 weeks-Month 3: number analyzed (Participants) | 12
  Tofacitinib monotherapy: < 6 weeks-Month 3 | 3
  Tofacitinib monotherapy: >= 6 weeks-Month 3: number analyzed (Participants) | 24
  Tofacitinib monotherapy: >= 6 weeks-Month 3 | 3
  Tofacitinib monotherapy: Missing-Month 3: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Missing-Month 3 | 2
  Tofacitinib monotherapy: < 6 weeks-Month 6: number analyzed (Participants) | 13
  Tofacitinib monotherapy: < 6 weeks-Month 6 | 7
  Tofacitinib monotherapy: >= 6 weeks-Month 6: number analyzed (Participants) | 13
  Tofacitinib monotherapy: >= 6 weeks-Month 6 | 7
  Tofacitinib monotherapy: Missing-Month 6: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Missing-Month 6 | 1
  Tofacitinib monotherapy: < 6 weeks-Month 12: number analyzed (Participants) | 9
  Tofacitinib monotherapy: < 6 weeks-Month 12 | 2
  Tofacitinib monotherapy: >= 6 weeks-Month 12: number analyzed (Participants) | 10
  Tofacitinib monotherapy: >= 6 weeks-Month 12 | 7
  Combined tofacitinib and MTX therapy: < 6 weeks-Month 3: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: < 6 weeks-Month 3 | 1
  Combined tofacitinib and MTX therapy: >= 6 weeks-Month 3: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: >= 6 weeks-Month 3 | 3
  Combined tofacitinib and MTX therapy: < 6 weeks-Month 6: number analyzed (Participants) | 6
  Combined tofacitinib and MTX therapy: < 6 weeks-Month 6 | 4
  Combined tofacitinib and MTX therapy: >= 6 weeks-Month 6: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: >= 6 weeks-Month 6 | 1
  Combined tofacitinib and MTX therapy: < 6 weeks-Month 12: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: < 6 weeks-Month 12 | 2
  Combined tofacitinib and MTX therapy: >= 6 weeks-Month 12: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: >= 6 weeks-Month 12 | 1
  Combined tofacitinib and other csDMARD: >= 6 weeks-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: >= 6 weeks-Month 3 | 0

11. Secondary Outcome: Number of Participants Who Achieved LDA According to Erythrocyte Sedimentation Rate (ESR) Results at Months 3, 6 and 12
Description: ESR result=abnormal if test result was above normal range. ESR normal range:0-50 years(male <15 mm/h, female <20 mm/h), 51-85 years(<20 mm/h males and <30 mm/h females),older than 85 years(<30 mm/h males and <42 mm/h females). Number of participants who achieved LDA according to ESR results(normal and abnormal) were reported. LDA=PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of following:participant global PAA,physician global PAA,each scored on 100 mm VAS,0=no DA, 100=maximum DA; TJC(0-68); SJC(0-66); LEI score=0-6;0=non tender,6=more enthesitis burden; tender dactylitis digit score=0-3,0=no tenderness,3=participant withdrew digit; PCS of SF-36 score=0-100; 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged=0(no disease)to 10(severe disease);higher scores=more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: Abnormal-Month 3: number analyzed (Participants) | 14
  Overall: Abnormal-Month 3 | 2
  Overall: Normal-Month 3: number analyzed (Participants) | 22
  Overall: Normal-Month 3 | 8
  Overall: Missing-Month 3: number analyzed (Participants) | 15
  Overall: Missing-Month 3 | 2
  Overall: Abnormal-Month 6: number analyzed (Participants) | 10
  Overall: Abnormal-Month 6 | 4
  Overall: Normal-Month 6: number analyzed (Participants) | 16
  Overall: Normal-Month 6 | 10
  Overall: Missing-Month 6: number analyzed (Participants) | 12
  Overall: Missing-Month 6 | 6
  Overall: Abnormal-Month 12: number analyzed (Participants) | 7
  Overall: Abnormal-Month 12 | 3
  Overall: Normal-Month 12: number analyzed (Participants) | 12
  Overall: Normal-Month 12 | 7
  Overall: Missing-Month 12: number analyzed (Participants) | 7
  Overall: Missing-Month 12 | 2
  Tofacitinib monotherapy: Abnormal-Month 3: number analyzed (Participants) | 8
  Tofacitinib monotherapy: Abnormal-Month 3 | 1
  Tofacitinib monotherapy: Normal-Month 3: number analyzed (Participants) | 17
  Tofacitinib monotherapy: Normal-Month 3 | 6
  Tofacitinib monotherapy: Missing-Month 3: number analyzed (Participants) | 13
  Tofacitinib monotherapy: Missing-Month 3 | 1
  Tofacitinib monotherapy: Abnormal-Month 6: number analyzed (Participants) | 6
  Tofacitinib monotherapy: Abnormal-Month 6 | 2
  Tofacitinib monotherapy: Normal-Month 6: number analyzed (Participants) | 11
  Tofacitinib monotherapy: Normal-Month 6 | 8
  Tofacitinib monotherapy: Missing-Month 6: number analyzed (Participants) | 10
  Tofacitinib monotherapy: Missing-Month 6 | 5
  Tofacitinib monotherapy: Abnormal-Month 12: number analyzed (Participants) | 4
  Tofacitinib monotherapy: Abnormal-Month 12 | 2
  Tofacitinib monotherapy: Normal-Month 12: number analyzed (Participants) | 10
  Tofacitinib monotherapy: Normal-Month 12 | 5
  Tofacitinib monotherapy: Missing-Month 12: number analyzed (Participants) | 5
  Tofacitinib monotherapy: Missing-Month 12 | 2
  Combined tofacitinib and MTX therapy: Abnormal-Month 3: number analyzed (Participants) | 6
  Combined tofacitinib and MTX therapy: Abnormal-Month 3 | 1
  Combined tofacitinib and MTX therapy: Normal-Month 3: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Normal-Month 3 | 2
  Combined tofacitinib and MTX therapy: Missing-Month 3: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: Missing-Month 3 | 1
  Combined tofacitinib and MTX therapy: Abnormal-Month 6: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Abnormal-Month 6 | 2
  Combined tofacitinib and MTX therapy: Normal-Month 6: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: Normal-Month 6 | 2
  Combined tofacitinib and MTX therapy: Missing-Month 6: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: Missing-Month 6 | 1
  Combined tofacitinib and MTX therapy: Abnormal-Month 12: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: Abnormal-Month 12 | 1
  Combined tofacitinib and MTX therapy: Normal-Month 12: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: Normal-Month 12 | 2
  Combined tofacitinib and MTX therapy: Missing-Month 12: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: Missing-Month 12 | 0
  Combined tofacitinib and other csDMARD: Normal-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Normal-Month 3 | 0

12. Secondary Outcome: Number of Participants Who Achieved LDA According to C-reactive Protein (CRP) Results at Months 3, 6 and 12
Description: For CRP, result was considered abnormal if t the test result was above the normal range (0.3 to 10 mg/L). LDA was defined as PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: Abnormal-Month 3: number analyzed (Participants) | 20
  Overall: Abnormal-Month 3 | 7
  Overall: Normal-Month 3: number analyzed (Participants) | 31
  Overall: Normal-Month 3 | 5
  Overall: Abnormal-Month 6: number analyzed (Participants) | 14
  Overall: Abnormal-Month 6 | 8
  Overall: Normal-Month 6: number analyzed (Participants) | 24
  Overall: Normal-Month 6 | 12
  Overall: Abnormal-Month 12: number analyzed (Participants) | 8
  Overall: Abnormal-Month 12 | 4
  Overall: Normal-Month 12: number analyzed (Participants) | 18
  Overall: Normal-Month 12 | 8
  Tofacitinib monotherapy: Abnormal-Month 3: number analyzed (Participants) | 15
  Tofacitinib monotherapy: Abnormal-Month 3 | 4
  Tofacitinib monotherapy: Normal-Month 3: number analyzed (Participants) | 23
  Tofacitinib monotherapy: Normal-Month 3 | 4
  Tofacitinib monotherapy: Abnormal-Month 6: number analyzed (Participants) | 10
  Tofacitinib monotherapy: Abnormal-Month 6 | 5
  Tofacitinib monotherapy: Normal-Month 6: number analyzed (Participants) | 17
  Tofacitinib monotherapy: Normal-Month 6 | 10
  Tofacitinib monotherapy: Abnormal-Month 12: number analyzed (Participants) | 4
  Tofacitinib monotherapy: Abnormal-Month 12 | 2
  Tofacitinib monotherapy: Normal-Month 12: number analyzed (Participants) | 15
  Tofacitinib monotherapy: Normal-Month 12 | 7
  Combined tofacitinib and MTX therapy: Abnormal-Month 3: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: Abnormal-Month 3 | 3
  Combined tofacitinib and MTX therapy: Normal-Month 3: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Normal-Month 3 | 1
  Combined tofacitinib and MTX therapy: Abnormal-Month 6: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Abnormal-Month 6 | 3
  Combined tofacitinib and MTX therapy: Normal-Month 6: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Normal-Month 6 | 2
  Combined tofacitinib and MTX therapy: Abnormal-Month 12: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Abnormal-Month 12 | 2
  Combined tofacitinib and MTX therapy: Normal-Month 12: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: Normal-Month 12 | 1
  Combined tofacitinib and other csDMARD: Normal-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Normal-Month 3 | 0

13. Secondary Outcome: Number of Participants Who Achieved LDA According to Presence of Rheumatoid Nodules at Months 3, 6 and 12
Description: Number of participants who achieved LDA according to presence (present/absent) of rheumatoid nodules is presented in this outcome measure. LDA was defined as PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: Absent-Month 3: number analyzed (Participants) | 49
  Overall: Absent-Month 3 | 12
  Overall: Missing-Month 3: number analyzed (Participants) | 2
  Overall: Missing-Month 3 | 0
  Overall: Absent-Month 6: number analyzed (Participants) | 37
  Overall: Absent-Month 6 | 20
  Overall: Missing-Month 6: number analyzed (Participants) | 1
  Overall: Missing-Month 6 | 0
  Overall: Absent-Month 12: number analyzed (Participants) | 25
  Overall: Absent-Month 12 | 12
  Overall: Missing-Month 12: number analyzed (Participants) | 1
  Overall: Missing-Month 12 | 0
  Tofacitinib monotherapy: Absent-Month 3: number analyzed (Participants) | 36
  Tofacitinib monotherapy: Absent-Month 3 | 8
  Tofacitinib monotherapy: Missing-Month 3: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Missing-Month 3 | 0
  Tofacitinib monotherapy: Absent-Month 6: number analyzed (Participants) | 26
  Tofacitinib monotherapy: Absent-Month 6 | 15
  Tofacitinib monotherapy: Missing-Month 6: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Missing-Month 6 | 0
  Tofacitinib monotherapy: Absent-Month 12: number analyzed (Participants) | 18
  Tofacitinib monotherapy: Absent-Month 12 | 9
  Tofacitinib monotherapy: Missing-Month 12: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Missing-Month 12 | 0
  Combined tofacitinib and MTX therapy: Absent-Month 3: number analyzed (Participants) | 12
  Combined tofacitinib and MTX therapy: Absent-Month 3 | 4
  Combined tofacitinib and MTX therapy: Absent-Month 6: number analyzed (Participants) | 11
  Combined tofacitinib and MTX therapy: Absent-Month 6 | 5
  Combined tofacitinib and MTX therapy: Absent-Month 12: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Absent-Month 12 | 3
  Combined tofacitinib and other csDMARD: Absent-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Absent-Month 3 | 0

14. Secondary Outcome: Number of Participants Who Achieved LDA According to Presence of Unequivocal Radiological Erosion at Months 3, 6 and 12
Description: Unequivocal radiological erosion: 'present',if Sharp-Van der Heijde modified score (S-VH MS)for erosion >0;'absent',if S-VH MS for erosion score=0. S-VH MS sum of erosion,JSN scores(range 0-528). Higher score=more severe disease. If a component score is missing, S-VH MS is missing. LDA=PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of following: participant global PAA,physician global PAA,each scored on 100 mm VAS,0=no DA,100=maximum DA; TJC(0-68); SJC(0-66); LEI score range=0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score range=0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score range=0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0(no disease)to 10(severe disease); higher scores=more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: Present-Month 3: number analyzed (Participants) | 2
  Overall: Present-Month 3 | 1
  Overall: Absent-Month 3: number analyzed (Participants) | 4
  Overall: Absent-Month 3 | 1
  Overall: Missing-Month 3: number analyzed (Participants) | 45
  Overall: Missing-Month 3 | 10
  Overall: Present-Month 6: number analyzed (Participants) | 1
  Overall: Present-Month 6 | 1
  Overall: Absent-Month 6: number analyzed (Participants) | 5
  Overall: Absent-Month 6 | 2
  Overall: Missing-Month 6: number analyzed (Participants) | 32
  Overall: Missing-Month 6 | 17
  Overall: Present-Month 12: number analyzed (Participants) | 1
  Overall: Present-Month 12 | 0
  Overall: Absent-Month 12: number analyzed (Participants) | 1
  Overall: Absent-Month 12 | 1
  Overall: Missing-Month 12: number analyzed (Participants) | 24
  Overall: Missing-Month 12 | 11
  Tofacitinib monotherapy: Present-Month 3: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Present-Month 3 | 1
  Tofacitinib monotherapy: Absent-Month 3: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Absent-Month 3 | 0
  Tofacitinib monotherapy: Missing-Month 3: number analyzed (Participants) | 35
  Tofacitinib monotherapy: Missing-Month 3 | 7
  Tofacitinib monotherapy: Present-Month 6: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Present-Month 6 | 1
  Tofacitinib monotherapy: Absent-Month 6: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Absent-Month 6 | 2
  Tofacitinib monotherapy: Missing-Month 6: number analyzed (Participants) | 24
  Tofacitinib monotherapy: Missing-Month 6 | 12
  Tofacitinib monotherapy: Present-Month 12: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Present-Month 12 | 0
  Tofacitinib monotherapy: Absent-Month 12: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Absent-Month 12 | 1
  Tofacitinib monotherapy: Missing-Month 12: number analyzed (Participants) | 17
  Tofacitinib monotherapy: Missing-Month 12 | 8
  Combined tofacitinib and MTX therapy: Absent-Month 3: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: Absent-Month 3 | 1
  Combined tofacitinib and MTX therapy: Missing-Month 3: number analyzed (Participants) | 9
  Combined tofacitinib and MTX therapy: Missing-Month 3 | 3
  Combined tofacitinib and MTX therapy: Absent-Month 6: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: Absent-Month 6 | 0
  Combined tofacitinib and MTX therapy: Missing-Month 6: number analyzed (Participants) | 8
  Combined tofacitinib and MTX therapy: Missing-Month 6 | 5
  Combined tofacitinib and MTX therapy: Missing-Month 12: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Missing-Month 12 | 3
  Combined tofacitinib and other csDMARD: Missing-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Missing-Month 3 | 0

15. Secondary Outcome: Number of Participants Who Achieved LDA According to Presence of Unequivocal Bony Decalcification Localized to the Joints of the Hands and Wrists at Months 3, 6 and 12
Description: Unequivocal Bony decalcification was reported as present or absent at enrollment. LDA was defined as PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of the following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: Present-Month 3: number analyzed (Participants) | 2
  Overall: Present-Month 3 | 1
  Overall: Absent-Month 3: number analyzed (Participants) | 38
  Overall: Absent-Month 3 | 7
  Overall: Missing-Month 3: number analyzed (Participants) | 11
  Overall: Missing-Month 3 | 4
  Overall: Present-Month 6: number analyzed (Participants) | 3
  Overall: Present-Month 6 | 3
  Overall: Absent-Month 6: number analyzed (Participants) | 27
  Overall: Absent-Month 6 | 12
  Overall: Missing-Month 6: number analyzed (Participants) | 8
  Overall: Missing-Month 6 | 5
  Overall: Present-Month 12: number analyzed (Participants) | 3
  Overall: Present-Month 12 | 2
  Overall: Absent-Month 12: number analyzed (Participants) | 16
  Overall: Absent-Month 12 | 7
  Overall: Missing-Month 12: number analyzed (Participants) | 7
  Overall: Missing-Month 12 | 3
  Tofacitinib monotherapy: Present-Month 3: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Present-Month 3 | 1
  Tofacitinib monotherapy: Absent-Month 3: number analyzed (Participants) | 30
  Tofacitinib monotherapy: Absent-Month 3 | 6
  Tofacitinib monotherapy: Missing-Month 3: number analyzed (Participants) | 7
  Tofacitinib monotherapy: Missing-Month 3 | 1
  Tofacitinib monotherapy: Present-Month 6: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Present-Month 6 | 2
  Tofacitinib monotherapy: Absent-Month 6: number analyzed (Participants) | 21
  Tofacitinib monotherapy: Absent-Month 6 | 11
  Tofacitinib monotherapy: Missing-Month 6: number analyzed (Participants) | 4
  Tofacitinib monotherapy: Missing-Month 6 | 2
  Tofacitinib monotherapy: Present-Month 12: number analyzed (Participants) | 2
  Tofacitinib monotherapy: Present-Month 12 | 1
  Tofacitinib monotherapy: Absent-Month 12: number analyzed (Participants) | 13
  Tofacitinib monotherapy: Absent-Month 12 | 6
  Tofacitinib monotherapy: Missing-Month 12: number analyzed (Participants) | 4
  Tofacitinib monotherapy: Missing-Month 12 | 2
  Combined tofacitinib and MTX therapy: Present-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: Present-Month 3 | 0
  Combined tofacitinib and MTX therapy: Absent-Month 3: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Absent-Month 3 | 1
  Combined tofacitinib and MTX therapy: Missing-Month 3: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Missing-Month 3 | 3
  Combined tofacitinib and MTX therapy: Present-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: Present-Month 6 | 1
  Combined tofacitinib and MTX therapy: Absent-Month 6: number analyzed (Participants) | 6
  Combined tofacitinib and MTX therapy: Absent-Month 6 | 1
  Combined tofacitinib and MTX therapy: Missing-Month 6: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Missing-Month 6 | 3
  Combined tofacitinib and MTX therapy: Present-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: Present-Month 12 | 1
  Combined tofacitinib and MTX therapy: Absent-Month 12: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: Absent-Month 12 | 1
  Combined tofacitinib and MTX therapy: Missing-Month 12: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: Missing-Month 12 | 1
  Combined tofacitinib and other csDMARD: Absent-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Absent-Month 3 | 0

16. Secondary Outcome: Number of Participants Who Achieved LDA According to Presence of Symmetric Arthritis at Months 3, 6 and 12
Description: Arthritis at enrollment was identified when a participant reported swelling and/or tenderness/pain in any joint. Number of participants who achieved LDA according to presence (Yes/No) of symmetric arthritis was reported. LDA was defined as PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of following: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC (0-68); SJC (0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: No-Month 3: number analyzed (Participants) | 49
  Overall: No-Month 3 | 12
  Overall: Yes-Month 3: number analyzed (Participants) | 2
  Overall: Yes-Month 3 | 0
  Overall: No-Month 6: number analyzed (Participants) | 37
  Overall: No-Month 6 | 20
  Overall: Yes-Month 6: number analyzed (Participants) | 1
  Overall: Yes-Month 6 | 0
  Overall: No-Month 12: number analyzed (Participants) | 26
  Overall: No-Month 12 | 12
  Tofacitinib monotherapy: No-Month 3: number analyzed (Participants) | 37
  Tofacitinib monotherapy: No-Month 3 | 8
  Tofacitinib monotherapy: Yes-Month 3: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Yes-Month 3 | 0
  Tofacitinib monotherapy: No-Month 6: number analyzed (Participants) | 26
  Tofacitinib monotherapy: No-Month 6 | 15
  Tofacitinib monotherapy: Yes-Month 6: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Yes-Month 6 | 0
  Tofacitinib monotherapy: No-Month 12: number analyzed (Participants) | 19
  Tofacitinib monotherapy: No-Month 12 | 9
  Combined tofacitinib and MTX therapy: No-Month 3: number analyzed (Participants) | 11
  Combined tofacitinib and MTX therapy: No-Month 3 | 4
  Combined tofacitinib and MTX therapy: Yes-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: Yes-Month 3 | 0
  Combined tofacitinib and MTX therapy: No-Month 6: number analyzed (Participants) | 11
  Combined tofacitinib and MTX therapy: No-Month 6 | 5
  Combined tofacitinib and MTX therapy: No-Month 12: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: No-Month 12 | 3
  Combined tofacitinib and other csDMARD: No-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: No-Month 3 | 0

17. Secondary Outcome: Number of Participants Who Achieved LDA According to Arthritis of the Hand Joints at Months 3, 6 and 12
Description: Hand joints included metacarpal phalangeal joints(MCP), finger proximal interphalangeal and finger distal interphalangeal joints. Number of participants who achieved LDA according to presence(Yes/No) of arthritis of any of hand joints was reported. LDA=PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA which incorporated assessment of following: participant global PAA,physician global PAA, each scored on 100 mm VAS,0=no DA,100=maximum DA;TJC(0-68); SJC(0-66); LEI score ranging from 0-6; where 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; where 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores indicated more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: No-Month 3: number analyzed (Participants) | 12
  Overall: No-Month 3 | 4
  Overall: Yes-Month 3: number analyzed (Participants) | 39
  Overall: Yes-Month 3 | 8
  Overall: No-Month 6: number analyzed (Participants) | 9
  Overall: No-Month 6 | 6
  Overall: Yes-Month 6: number analyzed (Participants) | 29
  Overall: Yes-Month 6 | 14
  Overall: No-Month 12: number analyzed (Participants) | 5
  Overall: No-Month 12 | 1
  Overall: Yes-Month 12: number analyzed (Participants) | 21
  Overall: Yes-Month 12 | 11
  Tofacitinib monotherapy: No-Month 3: number analyzed (Participants) | 8
  Tofacitinib monotherapy: No-Month 3 | 2
  Tofacitinib monotherapy: Yes-Month 3: number analyzed (Participants) | 30
  Tofacitinib monotherapy: Yes-Month 3 | 6
  Tofacitinib monotherapy: No-Month 6: number analyzed (Participants) | 5
  Tofacitinib monotherapy: No-Month 6 | 4
  Tofacitinib monotherapy: Yes-Month 6: number analyzed (Participants) | 22
  Tofacitinib monotherapy: Yes-Month 6 | 11
  Tofacitinib monotherapy: No-Month 12: number analyzed (Participants) | 2
  Tofacitinib monotherapy: No-Month 12 | 1
  Tofacitinib monotherapy: Yes-Month 12: number analyzed (Participants) | 17
  Tofacitinib monotherapy: Yes-Month 12 | 8
  Combined tofacitinib and MTX therapy: No-Month 3: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: No-Month 3 | 2
  Combined tofacitinib and MTX therapy: Yes-Month 3: number analyzed (Participants) | 8
  Combined tofacitinib and MTX therapy: Yes-Month 3 | 2
  Combined tofacitinib and MTX therapy: No-Month 6: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: No-Month 6 | 2
  Combined tofacitinib and MTX therapy: Yes-Month 6: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Yes-Month 6 | 3
  Combined tofacitinib and MTX therapy: No-Month 12: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: No-Month 12 | 0
  Combined tofacitinib and MTX therapy: Yes-Month 12: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Yes-Month 12 | 3
  Combined tofacitinib and other csDMARD: Yes-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Yes-Month 3 | 0

18. Secondary Outcome: Number of Participants Who Achieved LDA According to Arthritis of Only 1 Medium-Large Joint at Months 3, 6 and 12
Description: Medium joints=temporomandibular, sternoclavicular, acromioclavicular, finger proximal interphalangeal, finger distal interphalangeal and tarsus/midfoot(feet) joints. Large joints=glenohumeral, elbows, hips, knees and ankles joint. Number of participants who achieved LDA according to presence (Yes/No) of arthritis of only 1 medium-large joint was reported. LDA=PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA incorporated assessment of: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA;TJC(0-68);SJC(0-66); LEI score ranging from 0-6;0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3;0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100;0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS score (0-10) uses a weighted formula; higher scores=more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: No-Month 3: number analyzed (Participants) | 44
  Overall: No-Month 3 | 10
  Overall: Yes-Month 3: number analyzed (Participants) | 7
  Overall: Yes-Month 3 | 2
  Overall: No-Month 6: number analyzed (Participants) | 34
  Overall: No-Month 6 | 17
  Overall: Yes-Month 6: number analyzed (Participants) | 4
  Overall: Yes-Month 6 | 3
  Overall: No-Month 12: number analyzed (Participants) | 24
  Overall: No-Month 12 | 11
  Overall: Yes-Month 12: number analyzed (Participants) | 2
  Overall: Yes-Month 12 | 1
  Tofacitinib monotherapy: No-Month 3: number analyzed (Participants) | 33
  Tofacitinib monotherapy: No-Month 3 | 7
  Tofacitinib monotherapy: Yes-Month 3: number analyzed (Participants) | 5
  Tofacitinib monotherapy: Yes-Month 3 | 1
  Tofacitinib monotherapy: No-Month 6: number analyzed (Participants) | 26
  Tofacitinib monotherapy: No-Month 6 | 14
  Tofacitinib monotherapy: Yes-Month 6: number analyzed (Participants) | 1
  Tofacitinib monotherapy: Yes-Month 6 | 1
  Tofacitinib monotherapy: No-Month 12: number analyzed (Participants) | 19
  Tofacitinib monotherapy: No-Month 12 | 9
  Combined tofacitinib and MTX therapy: No-Month 3: number analyzed (Participants) | 10
  Combined tofacitinib and MTX therapy: No-Month 3 | 3
  Combined tofacitinib and MTX therapy: Yes-Month 3: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: Yes-Month 3 | 1
  Combined tofacitinib and MTX therapy: No-Month 6: number analyzed (Participants) | 8
  Combined tofacitinib and MTX therapy: No-Month 6 | 3
  Combined tofacitinib and MTX therapy: Yes-Month 6: number analyzed (Participants) | 3
  Combined tofacitinib and MTX therapy: Yes-Month 6 | 2
  Combined tofacitinib and MTX therapy: No-Month 12: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: No-Month 12 | 2
  Combined tofacitinib and MTX therapy: Yes-Month 12: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: Yes-Month 12 | 1
  Combined tofacitinib and other csDMARD: No-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: No-Month 3 | 0

19. Secondary Outcome: Number of Participants Who Achieved LDA According to Arthritis of 2-10 Medium-Large Joints and/or 1-3 Small Joints at Months 3, 6 and 12
Description: Medium joints=temporomandibular, sternoclavicular, acromioclavicular, finger proximal interphalangeal (IP), finger distal interphalangeal, tarsus/midfoot (feet). Large joints=glenohumeral, elbows, hips, knees, ankles. Small joints=MCP, proximal IP, second through fifth metatarsal phalangeal (MTP), thumb IP, wrists. Number of participants who achieved LDA according to presence (Yes/No) arthritis of 2-10 medium-large joints and/or 1-3 small joints was reported. LDA=PASDAS score =<3.2. PASDAS is a composite PsA activity score including: participant /physician global (VAS 0-100; 0=no DA, 100=maximum DA), TJC (0-68), SJC (0-66), LEI (0-6; 0=non tender, 6=more enthesitis burden), tender dactylitis digit score (0-3; 0=no tenderness, 3=participant withdrew digit), SF-36 PCS (0-100; 0=severe physical health limitations, 100=excellent physical health),CRP in mg/L. PASDAS score (0-10) uses a weighted formula; higher scores=more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: No-Month 3: number analyzed (Participants) | 1
  Overall: No-Month 3 | 0
  Overall: Yes-Month 3: number analyzed (Participants) | 50
  Overall: Yes-Month 3 | 12
  Overall: No-Month 6: number analyzed (Participants) | 1
  Overall: No-Month 6 | 1
  Overall: Yes-Month 6: number analyzed (Participants) | 37
  Overall: Yes-Month 6 | 19
  Overall: No-Month 12: number analyzed (Participants) | 1
  Overall: No-Month 12 | 1
  Overall: Yes-Month 12: number analyzed (Participants) | 25
  Overall: Yes-Month 12 | 11
  Tofacitinib monotherapy: No-Month 3: number analyzed (Participants) | 1
  Tofacitinib monotherapy: No-Month 3 | 0
  Tofacitinib monotherapy: Yes-Month 3: number analyzed (Participants) | 37
  Tofacitinib monotherapy: Yes-Month 3 | 8
  Tofacitinib monotherapy: No-Month 6: number analyzed (Participants) | 1
  Tofacitinib monotherapy: No-Month 6 | 1
  Tofacitinib monotherapy: Yes-Month 6: number analyzed (Participants) | 26
  Tofacitinib monotherapy: Yes-Month 6 | 14
  Tofacitinib monotherapy: No-Month 12: number analyzed (Participants) | 1
  Tofacitinib monotherapy: No-Month 12 | 1
  Tofacitinib monotherapy: Yes-Month 12: number analyzed (Participants) | 18
  Tofacitinib monotherapy: Yes-Month 12 | 8
  Combined tofacitinib and MTX therapy: Yes-Month 3: number analyzed (Participants) | 12
  Combined tofacitinib and MTX therapy: Yes-Month 3 | 4
  Combined tofacitinib and MTX therapy: Yes-Month 6: number analyzed (Participants) | 11
  Combined tofacitinib and MTX therapy: Yes-Month 6 | 5
  Combined tofacitinib and MTX therapy: Yes-Month 12: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: Yes-Month 12 | 3
  Combined tofacitinib and other csDMARD: Yes-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Yes-Month 3 | 0

20. Secondary Outcome: Number of Participants Who Achieved LDA According to Arthritis of 4-10 Small Joints With or Without Involvement of Large Joints at Months 3, 6 and 12
Description: Large joints=glenohumeral, elbows, hips, knees and ankles joint. Small joints=MCP, proximal IP, second through fifth MTP, thumb IP, wrists. Number of participants who achieved LDA according to presence (Yes/No) of arthritis of 4-10 small joints with or without involvement of large joints was reported. LDA=PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA incorporated assessment of: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA;TJC(0-68); SJC(0-66); LEI score range=0-6; 0=non tender, 6=more enthesitis burden; tender dactylitis digit score range=0-3; 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores=more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: No-Month 3: number analyzed (Participants) | 25
  Overall: No-Month 3 | 8
  Overall: Yes-Month 3: number analyzed (Participants) | 26
  Overall: Yes-Month 3 | 4
  Overall: No-Month 6: number analyzed (Participants) | 19
  Overall: No-Month 6 | 12
  Overall: Yes-Month 6: number analyzed (Participants) | 19
  Overall: Yes-Month 6 | 8
  Overall: No-Month 12: number analyzed (Participants) | 13
  Overall: No-Month 12 | 6
  Overall: Yes-Month 12: number analyzed (Participants) | 13
  Overall: Yes-Month 12 | 6
  Tofacitinib monotherapy: No-Month 3: number analyzed (Participants) | 17
  Tofacitinib monotherapy: No-Month 3 | 4
  Tofacitinib monotherapy: Yes-Month 3: number analyzed (Participants) | 21
  Tofacitinib monotherapy: Yes-Month 3 | 4
  Tofacitinib monotherapy: No-Month 6: number analyzed (Participants) | 12
  Tofacitinib monotherapy: No-Month 6 | 8
  Tofacitinib monotherapy: Yes-Month 6: number analyzed (Participants) | 15
  Tofacitinib monotherapy: Yes-Month 6 | 7
  Tofacitinib monotherapy: No-Month 12: number analyzed (Participants) | 8
  Tofacitinib monotherapy: No-Month 12 | 4
  Tofacitinib monotherapy: Yes-Month 12: number analyzed (Participants) | 11
  Tofacitinib monotherapy: Yes-Month 12 | 5
  Combined tofacitinib and MTX therapy: No-Month 3: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: No-Month 3 | 4
  Combined tofacitinib and MTX therapy: Yes-Month 3: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: Yes-Month 3 | 0
  Combined tofacitinib and MTX therapy: No-Month 6: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: No-Month 6 | 4
  Combined tofacitinib and MTX therapy: Yes-Month 6: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Yes-Month 6 | 1
  Combined tofacitinib and MTX therapy: No-Month 12: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: No-Month 12 | 2
  Combined tofacitinib and MTX therapy: Yes-Month 12: number analyzed (Participants) | 2
  Combined tofacitinib and MTX therapy: Yes-Month 12 | 1
  Combined tofacitinib and other csDMARD: No-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: No-Month 3 | 0

21. Secondary Outcome: Number of Participants Who Achieved LDA According to Arthritis of >10 Joints (With at Least One Small Joint) at Months 3, 6 and 12
Description: Small joints=MCP, proximal IP, second through fifth MTP, thumb IP, wrists. Number of participants who achieved LDA according to presence (Yes/No) of arthritis of >10 joints (with at least one small joint) was reported in this outcome measure. LDA=PASDAS score =<3.2. PASDAS=composite disease activity measure for PsA incorporated assessment of: participant global PAA, physician global PAA, each scored on 100 mm VAS, 0=no DA, 100=maximum DA; TJC(0-68); SJC(0-66); LEI score ranging from 0-6; 0=non tender, 6=more enthesitis burden; tender dactylitis digit score ranging from 0-3; 0=no tenderness, 3=participant withdrew digit; PCS of SF-36 score ranging from 0-100; 0=severe physical health limitations and 100=excellent physical health and CRP in mg/L. PASDAS total score was calculated using a weighted formula and ranged from 0 (no disease) to 10 (severe disease); higher scores=more severe disease.
Time Frame: At Month 3, Month 6 and Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  Overall: No-Month 3: number analyzed (Participants) | 29
  Overall: No-Month 3 | 10
  Overall: Yes-Month 3: number analyzed (Participants) | 22
  Overall: Yes-Month 3 | 2
  Overall: No-Month 6: number analyzed (Participants) | 23
  Overall: No-Month 6 | 16
  Overall: Yes-Month 6: number analyzed (Participants) | 15
  Overall: Yes-Month 6 | 4
  Overall: No-Month 12: number analyzed (Participants) | 18
  Overall: No-Month 12 | 10
  Overall: Yes-Month 12: number analyzed (Participants) | 8
  Overall: Yes-Month 12 | 2
  Tofacitinib monotherapy: No-Month 3: number analyzed (Participants) | 21
  Tofacitinib monotherapy: No-Month 3 | 6
  Tofacitinib monotherapy: Yes-Month 3: number analyzed (Participants) | 17
  Tofacitinib monotherapy: Yes-Month 3 | 2
  Tofacitinib monotherapy: No-Month 6: number analyzed (Participants) | 16
  Tofacitinib monotherapy: No-Month 6 | 11
  Tofacitinib monotherapy: Yes-Month 6: number analyzed (Participants) | 11
  Tofacitinib monotherapy: Yes-Month 6 | 4
  Tofacitinib monotherapy: No-Month 12: number analyzed (Participants) | 12
  Tofacitinib monotherapy: No-Month 12 | 7
  Tofacitinib monotherapy: Yes-Month 12: number analyzed (Participants) | 7
  Tofacitinib monotherapy: Yes-Month 12 | 2
  Combined tofacitinib and MTX therapy: No-Month 3: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: No-Month 3 | 4
  Combined tofacitinib and MTX therapy: Yes-Month 3: number analyzed (Participants) | 5
  Combined tofacitinib and MTX therapy: Yes-Month 3 | 0
  Combined tofacitinib and MTX therapy: No-Month 6: number analyzed (Participants) | 7
  Combined tofacitinib and MTX therapy: No-Month 6 | 5
  Combined tofacitinib and MTX therapy: Yes-Month 6: number analyzed (Participants) | 4
  Combined tofacitinib and MTX therapy: Yes-Month 6 | 0
  Combined tofacitinib and MTX therapy: No-Month 12: number analyzed (Participants) | 6
  Combined tofacitinib and MTX therapy: No-Month 12 | 3
  Combined tofacitinib and MTX therapy: Yes-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and MTX therapy: Yes-Month 12 | 0
  Combined tofacitinib and other csDMARD: No-Month 3: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: No-Month 3 | 0

22. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Based on Short Form 36 (SF-36) Score at Months 3, 6 and 12
Description: The SF-36 is a participant administered scale assessing general quality of life. It consists of self-administered 36-item questionnaire that measured 8 health domains: physical function, role-physical, bodily pain, general health, vitality, social function, role-emotional, and mental health. These 8 domains are also summarized as physical and mental component scores. The score for each domain and component score is the mean of the individual question scores, which are scaled from 0 (minimum) to 100 (maximum), where high scores in each dimension and high overall scores indicate a better quality of life.
Time Frame: Baseline (measurement at enrollment), Month 3, Month 6 and Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 87
Units on a scale
  Overall: Physical health component summary score-Month 3 | 4.8 [3.00 to 6.56]
  Overall: Mental health component summary score-Month 3 | 2.4 [0.31 to 4.52]
  Tofacitinib monotherapy: Physical health component summary score-Month 3: number analyzed (Participants) | 64
  Tofacitinib monotherapy: Physical health component summary score-Month 3 | 5.0 [2.78 to 7.20]
  Tofacitinib monotherapy: Mental health component summary score-Month 3: number analyzed (Participants) | 64
  Tofacitinib monotherapy: Mental health component summary score-Month 3 | 2.5 [-0.23 to 5.26]
  Combined tofacitinib and MTX therapy: Physical health component summary score-Month 3: number analyzed (Participants) | 20
  Combined tofacitinib and MTX therapy: Physical health component summary score-Month 3 | 3.6 [0.67 to 6.44]
  Combined tofacitinib and MTX therapy: Mental health component summary score-Month 3: number analyzed (Participants) | 20
  Combined tofacitinib and MTX therapy: Mental health component summary score-Month 3 | 1.5 [-1.44 to 4.51]
  Combined tofacitinib and other csDMARD: Physical health component summary score-Month 3: number analyzed (Participants) | 3
  Combined tofacitinib and other csDMARD: Physical health component summary score-Month 3 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Combined tofacitinib and other csDMARD: Mental health component summary score-Month 3: number analyzed (Participants) | 3
  Combined tofacitinib and other csDMARD: Mental health component summary score-Month 3 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Overall: Physical health component summary score-Month 6: number analyzed (Participants) | 69
  Overall: Physical health component summary score-Month 6 | 5.5 [3.53 to 7.40]
  Overall: Mental health component summary score-Month 6: number analyzed (Participants) | 69
  Overall: Mental health component summary score-Month 6 | 2.6 [0.05 to 5.20]
  Tofacitinib monotherapy: Physical health component summary score-Month 6: number analyzed (Participants) | 49
  Tofacitinib monotherapy: Physical health component summary score-Month 6 | 6.2 [3.94 to 8.51]
  Tofacitinib monotherapy: Mental health component summary score-Month 6: number analyzed (Participants) | 49
  Tofacitinib monotherapy: Mental health component summary score-Month 6 | 2.9 [-0.41 to 6.20]
  Combined tofacitinib and MTX therapy: Physical health component summary score-Month 6: number analyzed (Participants) | 19
  Combined tofacitinib and MTX therapy: Physical health component summary score-Month 6 | 3.2 [-0.48 to 6.92]
  Combined tofacitinib and MTX therapy: Mental health component summary score-Month 6: number analyzed (Participants) | 19
  Combined tofacitinib and MTX therapy: Mental health component summary score-Month 6 | 0.9 [-3.22 to 5.01]
  Combined tofacitinib and other csDMARD: Physical health component summary score-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Physical health component summary score-Month 6 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Combined tofacitinib and other csDMARD: Mental health component summary score-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Mental health component summary score-Month 6 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Overall: Physical health component summary score-Month 12: number analyzed (Participants) | 55
  Overall: Physical health component summary score-Month 12 | 5.5 [3.33 to 7.69]
  Overall: Mental health component summary score-Month 12: number analyzed (Participants) | 55
  Overall: Mental health component summary score-Month 12 | 3.0 [0.11 to 5.83]
  Tofacitinib monotherapy: Physical health component summary score-Month 12: number analyzed (Participants) | 40
  Tofacitinib monotherapy: Physical health component summary score-Month 12 | 6.8 [4.06 to 9.45]
  Tofacitinib monotherapy: Mental health component summary score-Month 12: number analyzed (Participants) | 40
  Tofacitinib monotherapy: Mental health component summary score-Month 12 | 4.5 [1.04 to 8.03]
  Combined tofacitinib and MTX therapy: Physical health component summary score-Month 12: number analyzed (Participants) | 14
  Combined tofacitinib and MTX therapy: Physical health component summary score-Month 12 | 3.8 [0.60 to 6.97]
  Combined tofacitinib and MTX therapy: Mental health component summary score-Month 12: number analyzed (Participants) | 14
  Combined tofacitinib and MTX therapy: Mental health component summary score-Month 12 | -1.8 [-6.33 to 2.74]
  Combined tofacitinib and other csDMARD: Physical health component summary score-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Physical health component summary score-Month 12 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Combined tofacitinib and other csDMARD: Mental health component summary score-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD: Mental health component summary score-Month 12 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.

23. Secondary Outcome: Change From Baseline in QoL Based on Health Assessment Questionnaire - Disability Index (HAQ-DI41) at Months 3, 6 and 12
Description: The HAQ-DI41 assessed the degree of difficulty a participant had experienced during the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consisted of 2-3 items. For each question in the questionnaire, the level of difficulty was scored from 0 to 3 with 0 =no difficulty," 1 = "some difficulty," 2 = "much difficulty," and 3 = "unable to do". The disability index was computed by adding the scores for each of the components and dividing by the number of components with an available score. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: Baseline (measurement at enrollment), Month 3, Month 6 and Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 88
Units on a scale
  Overall-Month 3 | -0.1 [-0.21 to -0.01]
  Tofacitinib monotherapy-Month 3: number analyzed (Participants) | 64
  Tofacitinib monotherapy-Month 3 | -0.1 [-0.24 to 0.00]
  Combined tofacitinib and MTX therapy-Month 3: number analyzed (Participants) | 21
  Combined tofacitinib and MTX therapy-Month 3 | -0.0 [-0.23 to 0.14]
  Combined tofacitinib and other csDMARD-Month 3: number analyzed (Participants) | 3
  Combined tofacitinib and other csDMARD-Month 3 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Overall-Month 6: number analyzed (Participants) | 69
  Overall-Month 6 | -0.1 [-0.23 to 0.00]
  Tofacitinib monotherapy-Month 6: number analyzed (Participants) | 49
  Tofacitinib monotherapy-Month 6 | -0.1 [-0.29 to 0.01]
  Combined tofacitinib and MTX therapy-Month 6: number analyzed (Participants) | 19
  Combined tofacitinib and MTX therapy-Month 6 | 0.0 [-0.20 to 0.20]
  Combined tofacitinib and other csDMARD-Month 6: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 6 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.
  Overall-Month 12: number analyzed (Participants) | 54
  Overall-Month 12 | -0.2 [-0.32 to -0.02]
  Tofacitinib monotherapy-Month 12: number analyzed (Participants) | 39
  Tofacitinib monotherapy-Month 12 | -0.2 [-0.39 to -0.00]
  Combined tofacitinib and MTX therapy-Month 12: number analyzed (Participants) | 14
  Combined tofacitinib and MTX therapy-Month 12 | -0.2 [-0.39 to 0.07]
  Combined tofacitinib and other csDMARD-Month 12: number analyzed (Participants) | 1
  Combined tofacitinib and other csDMARD-Month 12 | NA [NA to NA] — Least squares mean and 95% CI limits could not be calculated due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: From Baseline (enrollment) until Month 12
Description: Same event may occur as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. SAF included all participants who received at least one dose (including partial dose) of study medication independently of inclusion/exclusion criteria.
Groups:
- All Participants: All participants with a diagnosis of PsA who received tofacitinib up to 12 months of follow-up were included in this retrospective observational study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/113
Serious Adverse Events (participants affected / at risk) | 7/113
Other Adverse Events (participants affected / at risk) | 50/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=113)
Pyelonephritis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=113)
Drug ineffective (General disorders) | 21
COVID-19 (Infections and infestations) | 10
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT04517669/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT04517669/SAP_001.pdf